CLINICAL TRIAL: NCT00910767
Title: A Randomised, 2-period Cross-over Study to Assess the Feasibility of Overnight Computer-based Glucose Control Based on Continuous Subcutaneous Glucose Monitoring, and Compare it With Conventional Pump Therapy in Adults With Type 1 Diabetes
Brief Title: Closing the Loop in Adults With Type 1 Diabetes
Acronym: ANGELA01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Diabetes UK (Other)
Responsible Party: Dr Mark Evans, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08/H0308/297
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed loop (algorithm) (Experimental)
  Interventions: Device: Closed loop
- Open loop (Placebo Comparator)
  Interventions: Device: Conventional insulin pump delivery

INTERVENTIONS:
Device: Conventional insulin pump delivery — Subcutaneous delivery of Novorapid insulin according to usual pump regime
  Arms: Open loop
Device: Closed loop — Subcutaneous delivery of Novorapid insulin, dose calculated by control algorithm, based on continuous glucose sensor readings
  Arms: Closed loop (algorithm)

SUMMARY:
The main objective of this study is to evaluate the feasibility of closed loop insulin pump therapy to improve overnight glucose control in adults with type 1 diabetes.

DETAILED DESCRIPTION:
People with type 1 diabetes(T1D) need regular insulin injections or continuous delivery of insulin using an insulin pump in order to keep the blood glucose levels normal. We know that keeping blood sugars in the normal range will help prevent long term diabetes related complications involving the eyes, kidneys and heart. However, achieving treatment goals can be very difficult as the tighter we try to control blood glucose levels, the greater the risk of the person developing episodes of low glucose levels (hypoglycaemia). This is a particular problem at night and one solution is to develop a system whereby the amount of insulin injected is very closely matched to the blood sugar levels on a continuous basis. This can be achieved by what is called a "closed loop system" where a small glucose sensor placed under the skin communicates with a computer containing an algorithm that drives an insulin pump. This system is being developed in Cambridge and we have trialed this on 16 children and adolescents with T1D in a clinical setting over the past year. We have found that this system is very effective at preventing hypoglycaemia in this group of patients.

We will recruit 12 adults with T1D on insulin pump therapy, and the studies will be done in a clinical research facility. The subjects will be studied on two nights. On one night they will have their normal insulin pump therapy and on the other night their insulin pump will be varied according to information about blood glucose values from the continuous glucose sensor. This information will be manually typed into the computer every 15 minutes from 8pm until 8am. The algorithm will advise of the insulin infusion rate and this will be manually changed by a trained nurse every 15 minutes throughout the night.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes, as defined by WHO for at least 6 months or confirmed C-peptide negative.
* On insulin pump therapy for at least 3 months

Exclusion Criteria:

* Non-type 1 diabetes mellitus
* Any physical/psychological disease likely to interfere with the study
* Taking medication likely to interfere with interpretation of the results
* Known/suspected allergy against insulin
* Patients with clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator
* Ongoing severe recurrent hypoglycaemia as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percentage of plasma glucose values in target (3.9 - 8.0 mmol/L) | 1900 to 0800hr

SECONDARY OUTCOMES:
Percentage of CGM (continuous glucose monitoring) values in target (3.9-8.0 mmol/L) | 1900 to 0800hr
Percentage of plasma glucose and CGM values in target (3.9-8.0 mmol/L) | 0000 to 0800hr
Percentage of plasma glucose and CGM values in target (3.9-8.0 mmol/L) | 0800 to 1200hr
Percentage of plasma glucose and CGM values below 3.9 mmol/L | 1900 to 0800hr
Percentage of plasma glucose and CGM values below 3.9 mmol/L | 0000 to 0800hr
Percentage of plasma glucose and CGM values below 3.9 mmol/L | 0800 to 1200hr
Percentage of plasma glucose and CGM values above 8.0 mmol/L | 1900 to 0800hr
Percentage of plasma glucose and CGM values above 8.0 mmol/L | 0000 to 0800hr
Percentage of plasma glucose and CGM values above 8.0 mmol/L | 0800 to 1200hr
Average plasma and CGM glucose | 1900 to 0800hr
Average plasma and CGM glucose | 0000 to 0800hr
Average plasma and CGM glucose | 0800 to 1200hr
Average plasma insulin concentration | 1900 to 0800hr
Average plasma insulin concentration | 0000 to 0800hr
Average plasma insulin concentration | 0800 to 1200hr
Total dose of insulin administered | 1900 to 0800hr
low blood glucose index (LBGI) score | 1900 to 0800hr
high blood glucose index (HBGI) score | 1900 to 0800hr
low blood glucose index (LBGI) score | 0000 to 0800hr
low blood glucose index (LBGI) score | 0800 to 1200hr
high blood glucose index (HBGI) score | 0000 to 0800hr
high blood glucose index (HBGI) score | 0800 to 1200hr
Percentage of plasma glucose and CGM values below 3.0 mmol/L | 1900 to 0800hr
Percentage of plasma glucose and CGM values below 3.0 mmol/L | 0000 to 0800hr
Percentage of plasma glucose and CGM values below 3.0 mmol/L | 0800 to 1200hr

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Evans, MD FRCP, Principal Investigator — University of Cambridge, UK; Roman Hovorka, PhD, Study Director — University of Cambridge, UK
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Hovorka R, Kumareswaran K, Harris J, Allen JM, Elleri D, Xing D, Kollman C, Nodale M, Murphy HR, Dunger DB, Amiel SA, Heller SR, Wilinska ME, Evans ML. Overnight closed loop insulin delivery (artificial pancreas) in adults with type 1 diabetes: crossover randomised controlled studies. BMJ. 2011 Apr 13;342:d1855. doi: 10.1136/bmj.d1855. PMID 21493665